CLINICAL TRIAL: NCT05601232
Title: A Phase II Study of Boron Neutron Capture Therapy (BNCT) for Patients With Unresectable Angiosarcoma, by Using CICS-1 and SPM-011
Brief Title: A Phase II Study by Using CICS-1 and SPM-011 Commissioned by CICS and STELLA PHARMA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stella Pharma Corporation (Industry)
Collaborators: Cancer Intelligence Care Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNCT-002/SPM-011-JAM002
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Unresectable Angiosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Boron Neutron Capture Therapy (BNCT) (Experimental)
  Interventions: Radiation: BNCT

INTERVENTIONS:
Radiation: BNCT — Patients will be infused SPM-011 intravenously at a dose of 200mg/kg/hr over 2 hours. Thereafter, patient will be infused SPM-011 intravenously at a dose of 100mg/kg/hr and will receive neutron irradiation simultaneously for a certain period of time based on his Boronophenylalanine (BPA) concentration in the blood.

SUMMARY:
The purpose of the study is to investigate efficacy and safety Boron Neutron Capture Therapy (BNCT) by using CICS-1 accelerator-based neutron capture therapy device with lithium targets developed by CICS, and the SPM-011 boron compound for use in BNCT developed by STELLA PHARMA in the treatment of unresectable angiosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained from the subject.
* Histologically documented primary skin angiosarcoma.
* Locally advanced or locally recurrent angiosarcoma, and not eligible for curative surgery, chemoradiotherapy or radiotherapy. (Including cases where the individual refuses treatment.)
* Measurable disease, as defined by RECIST v1.1.
* The longest diameter of the entire target lesion is 15 cm or less.
* ECOG performance status score of Grade 0 to 2

Exclusion Criteria:

* Apparent disseminated tumor lesions.
* Hereditary fructose intolerance.
* Phenylketonuria.
* Any serious concomitant disease that precludes completion of the study treatment.
* The target lesion has received radiation exceeding 75 Gy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Response rate as assessed by the Independent Review Facility (IRF) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Baseline until Day90
  Percentage of patients with response (CR or PR) for target lesions within 90 days after BNCT

SECONDARY OUTCOMES:
Response rate as assessed by the investigator according to RECISTv1.1 | Baseline until Day90
  Percentage of patients with response (CR or PR) for target lesions within 90 days after BNCT
Duration of response as assessed by the IRF and the investigator | Baseline until disease progression or death
  From the initial occurrence of confirmed CR or PR for target lesions, whichever occurred at first, until confirmed disease progression or death, whichever occurred first
Time to response as assessed by the IRF | Baseline until the initial occurrence of CR or PR
  From the date of BNCT until the initial occurrence of confirmed CR or PR for target lesions, whichever occurred at first
Complete response (CR) rate as assessed by the IRF and the investigator | Baseline until the initial occurrence of CR
  Percentage of patients with CR for target lesions after BNCT
Disease control rate as assessed by the IRF and the investigator | Baseline until the initial occurrence of CR, PR or SD
  Percentage of patients with CR, PR and SD for target lesions after BNCT
Overall response rate as assessed by the IRF and the investigator | Baseline until the initial occurrence of CR or PR
  Percentage of patients with CR or PR after BNCT
Locoregional progression-free survival as assessed by the investigator | Baseline until in-field disease progression
  From the date of BNCT until confirmed in-field disease progression
Extra-regional relapse-free survival as assessed by the investigator | Baseline until extra-field disease progression
  From the date of BNCT until confirmed extra-field disease progression (new lesions)
Progression-free survival as assessed by the IRF and the investigator | Baseline until disease progression or death
  From the date of BNCT until confirmed disease progression or death, whichever occurred first
Maximum percent change in sum of tumor diameters of target lesions as assessed by the IRF and the investigator | Baseline until Day90
  Maximum percent change in sum of tumor diameters of target lesions within 90 days after BNCT
Overall survival | Baseline until death
  From the date of BNCT until death from any causes

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No